CLINICAL TRIAL: NCT01282723
Title: Multi-Reader Multi-Case Study to Identify Uterine Contractions Recorded From Laboring Patients by Practicing Clinicians
Status: Completed | Type: Observational
Sponsor: Reproductive Research Technologies, LP (Industry)
Responsible Party: Jack McCrary, Managing Director, Reproductive Research Technologies, LP
Other Study IDs: RRT-10-01
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-02

CONDITIONS: Pregnancy - Labor Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Pregnant, In Labor

SUMMARY:
This multi-reader multi-case study was designed to evaluate the performance of SureCALL® EMG Labor Monitor® (SureCALL®)to the predicate Tocodynamometer device (TOCO) using the performance of an Intrauterine Pressure Catheter device (IUPC) as the "gold standard".

DETAILED DESCRIPTION:
The SureCALL® EMG Labor Monitor® (SureCALL®)is a transabdominal electromyography monitor intended to measure intrapartum uterine activity. It is intended for use on term pregnant women who are in labor, with singleton pregnancies, using surface electrodes on the maternal abdomen. The device is intended for use by healthcare professionals in a clinical setting.

This multi-reader multi-case study was designed to evaluate the performance of SureCALL® to the predicate Tocodynamometer device (TOCO) using the performance of an Intrauterine Pressure Catheter device (IUPC) as the "gold standard".

This study involved 20 women at term, in labor, at three clinical sites. Each study subject was instrumented with three technologies for measuring uterine activity:

1. a tocodynamometer attached to the maternal abdomen
2. a set of abdominal surface electrodes for uterine electromyography, and
3. an intrauterine pressure catheter.

An assessment was obtained and quantified from masked, qualified clinical obstetrician readers for the evaluation of the equivalence of the three independent labor monitor devices by identifying in isolation the individual uterine contraction signals and the peak of each contraction signal produced by a full-term patient in term labor as independently collected by each labor monitor device.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy
* Indicated for IUPC
* Gestational ages from 37 to 41 weeks
* Informed consent required

Exclusion Criteria:

* Multifetal pregnancy
* Not Indicated for IUPC
* Gestation age below 37 or above 41 weeks
* Informed consent not given

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women in labor with uncomplicated singleton pregnancies and IUPC indicated with membranes ruptured and sufficient cervical dilation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Waterhouse, MD, Principal Investigator — Reproductive Research Technologies, LP
Locations (3):
- United States (3):
  - St.Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant, In Labor: Monitored simultaneously by SureCALL®, TOCO, and IUPC
Period: Overall Study
Arm/Group | Pregnant, In Labor
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant, In Labor
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 18
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.85 (4.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Comparison of SureCALL® and TOCO Detection of Contraction Events, as Compared to the IUPC, as Identified by Readers
Description: The presence of contractions measured by the SureCALL®, the presence of contractions measured by the TOCO, and the presence of contractions measured by the IUPC were determined by independent Readers. The Odds Ratio of SureCALL® contractions to IUPC contractions was calculated, and the Odd Ratio of TOCO contractions to IUPC contractions was calculated. Reader Correspondence was determined by a General Linear Mixed Model.
Time Frame: 9 - 42 Minutes
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Pregnant, In Labor
Number analyzed (Participants) | 20
Odds Ratio
  True Positive Fraction | 1.47 [1.10 to 1.95]
  False Positive Fraction | 0.85 [0.61 to 1.17]
Statistical Analysis 1: Comparison: Pregnant, In Labor; Estimation of Odds Ratio of True Positive Fraction between SureCALL® and TOCO Null hypothesis: There is no difference between the True Positive Fraction of SureCALL® and of TOCO or the SureCALL® is significantly greater than TOCO. Alternative hypothesis: There is a difference between the True Positive Fraction of SureCALL® and of TOCO and the TOCO is significantly greater than SureCALL®; Test type: Superiority or Other; p = 0.0093, Mixed Models Analysis; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.10 to 1.95]
Statistical Analysis 2: Comparison: Pregnant, In Labor; Estimation of Odds Ratio of False Positive Fraction between SureCALL® and TOCO Null hypothesis: There is no difference between the False Positive Fraction of SureCALL® and of TOCO or the SureCALL® is significantly less than TOCO. Alternative hypothesis: There is a difference between the False Positive Fraction of SureCALL® and of TOCO and the TOCO is significantly less than SureCALL®; Test type: Superiority or Other; p = 0.3204, Mixed Models Analysis; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.61 to 1.17]

ADVERSE EVENTS:
Arm/Group | Pregnant, In Labor
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may publish or present results of the study after the expiration of 12 months from completion. Publications or presentations are subject to the protection of confidential information or patentable information.